CLINICAL TRIAL: NCT07377890
Title: Accuracy of Intraorally Scanned Denture Impressions Compared to Conventional Border-Molded Impressions: An In Vivo Study
Brief Title: Accuracy of Digital vs Conventional Denture Impressions: An In Vivo Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Fatemeh Amir-Rad, Assistant Professor, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBRU IRB-2024-107
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Edentulism; Complete Dentures; Digital Impression Accuracy; Dental Impression Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Edentulous patients (Experimental): Arm Description:
  Participants will first receive digital intraoral scanning of their fully edentulous upper and/or lower jaw using the TRIOS 5 intraoral scanner (3Shape). The scanning process follows a structured sequence to capture the entire arch, including the palate and ridge slopes. Each arch will be scanned three times during the same visit to assess precision (consistency of repeated scans). Then the same participants will also undergo a conventional impression procedure using a custom tray and border molding technique.
  Interventions: Procedure: Digital and conventional impressions

INTERVENTIONS:
Procedure: Digital and conventional impressions — Participants will first receive digital intraoral scanning of their fully edentulous upper and/or lower jaw using the TRIOS 5 intraoral scanner (3Shape). The scanning process follows a structured sequence to capture the entire arch, including the palate and ridge slopes. Each arch will be scanned three times during the same visit to assess precision (consistency of repeated scans). Then the same participants will also undergo a conventional impression procedure using a custom tray and border molding technique.
  Other Names: intra-oral scanning; border-molded impression

SUMMARY:
The goal of this clinical trial is to compare the accuracy of two denture impression techniques, digital intraoral scanning and conventional border-molded impressions, in adults who have lost all their teeth (fully edentulous patients).

The main questions it aims to answer are:

Is a digital intraoral scan as accurate as a conventional impression for capturing the shape of the mouth, including movable gum areas? Are repeated digital scans consistent (precise) when taken multiple times on the same patient? Researchers will compare digital impressions taken with an intraoral scanner to conventional impressions made with custom trays and border molding to see if digital scans can match the accuracy of the traditional "gold standard" method.

Participants will:

Attend Dubai Dental Hospital for two study visits. Have their mouth scanned three times using a digital intraoral scanner. Have a conventional impression taken using a custom tray and high-accuracy material after border molding.

Provide informed consent and allow their impression data to be analyzed for accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending DDH for complete dental prosthesis.
* Fully edentulous patients
* All alveolar ridge classifications of Cawood and Howell 1988 (Cawood and Howell, 1988)
* Above 18 years old
* Arabic and English-speaking patients
* Good physical health (ASA class 1 or 2)
* Willing to provide informed consent.

Exclusion Criteria:

* Dentate patients
* Implant-attachment-supported complete denture.
* Patients un-willing to participate (non-consented patients)
* Patients with severe gag reflex
* Patients who are mentally unstable, drug users or alcoholics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Trueness of Digital Impressions: Mean root mean square Deviation (mm) between intraoral scanner (IOS) digital impressions and conventional impression scans-per arch | 1 week
  Trueness will be checked by looking at the Root Mean Square (RMS) deviation (mm) after superimposing the IOS Standard Tessellation Language (STL) over the conventional impression scan STL (reference) using Geomagic Control X. The primary metric is the participant-level mean RMS over the full arch surface (edentulous maxilla and mandible analyzed separately). Lower RMS indicates greater trueness (higher accuracy). Region-specific RMS (static vs. dynamic tissues) will be recorded as prespecified analyses (see secondary outcomes).
  Alignment: Initial + best-fit alignment; conventional scan = reference file. Reporting (participant level): Mean RMS (mm) per arch. Reporting (study level): Mean [Standard Deviation (SD)], RMS per arch; 95% CI; distribution plots as applicable.
  Unit of Measure: millimeters (mm), RMS deviation Regions analyzed: Static (palatal rugae, ridge slopes, crest) and dynamic (labial, buccal, lingual sulci, hamular notch, posterior palatal seal).
Precision of Digital Impressions: Within-Subject Mean Pairwise RMS Deviation (mm) Across Three IOS Scans (Precision)-per Arch | 1 week
  Precision will be quantified by pairwise deviation analysis between three repeated IOS scans per arch taken on the same day. STL files will be aligned (Initial + Best-Fit ICP) in Geomagic Control X. For each arch, the following pairs will be analyzed: (Scan1-Scan2), (Scan1-Scan3), and (Scan2-Scan3). Each pair will be aligned in both directions (each file alternately as reference), and all RMS values will be averaged to yield the participant-level mean pairwise RMS (mm) for that arch. Lower RMS indicates greater precision (repeatability).
  Reporting (participant level): Mean of all pairwise RMS values per arch. Reporting (study level): Mean (SD) RMS per arch; 95% CI; distribution plots as applicable.
  Unit of Measure: millimeters (mm), RMS deviation

SECONDARY OUTCOMES:
The difference (mm) in mean RMS trueness between the maxillary and mandibular arches is measured. | 1 week
  Compute mean RMS trueness (mm) per arch (as defined in Primary Outcome 1). The between-arch difference will be calculated as maxilla minus mandible (mm). Positive values indicate higher RMS (worse trueness) in the maxilla.
  Reporting (study level): Mean (SD) difference; 95% CI; paired analysis. Unit of Measure: millimeters (mm), RMS deviation
Difference (mm) in mean RMS trueness between static (attached) and dynamic (mobile) regions. | 1 week
  Within each arch, participant-level trueness RMS (mm) will be computed separately for prespecified static regions (palatal rugae; buccal and palatal/lingual slopes; ridge crest) and dynamic regions (labial, buccal, and lingual sulci; hamular notch; posterior palatal seal). The regional difference will be calculated as Dynamic minus Static (mm). Positive values indicate higher RMS (worse trueness) in mobile tissues.
  Reporting (study level): Mean (SD) difference; 95% CI; by arch as applicable. Unit of Measure: millimeters (mm), RMS deviation

OTHER OUTCOMES:
Difference (mm) in mean RMS precision between static (attached) and dynamic (mobile) regions. | 1 week
  Using the precision pipeline (Primary Outcome 2), compute regional mean pairwise RMS (mm) for static and dynamic regions per arch and participant, then calculate Dynamic minus Static (mm). Positive values indicate higher RMS (worse precision) in mobile tissues.
  Reporting (study level): Mean (SD) difference; 95% CI; by arch as applicable. Unit of Measure: millimeters (mm), RMS deviation

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Dental Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zarone F, Ruggiero G, Ferrari M, Mangano F, Joda T, Sorrentino R. Comparison of different intraoral scanning techniques on the completely edentulous maxilla: An in vitro 3-dimensional comparative analysis. J Prosthet Dent. 2020 Dec;124(6):762.e1-762.e8. doi: 10.1016/j.prosdent.2020.07.017. Epub 2020 Oct 24. PMID 33289648
- [Background] Al Hamad KQ, Al-Kaff FT. Trueness of intraoral scanning of edentulous arches: A comparative clinical study. J Prosthodont. 2023 Jan;32(1):26-31. doi: 10.1111/jopr.13597. Epub 2022 Sep 6. PMID 35997079
- [Background] Casucci A, Mazzitelli C, Tsiplakis V, D'Arienzo LF, Breschi L, Ferrari M. Digital Impressions in Edentulous Patients: A Systematic Review for Clinical Evidence. Int J Prosthodont. 2023 Sep 12;36(4):486-497. doi: 10.11607/ijp.7483. PMID 37699190
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35997079/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37699190/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33289648/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT07377890/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT07377890/ICF_001.pdf